CLINICAL TRIAL: NCT06212115
Title: The Effect of Donor-oriented Anti-infection Therapy Based on mNGS Etiological Diagnosis on the Incidence of Perioperative Infection and Prognosis of Corresponding Recipients After Liver Transplantation
Brief Title: Anti-infection Therapy Based on mNGS Etiological Diagnosis and Infection After Liver Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Shenzhen Third People's Hospital (Other)
Responsible Party: Principal Investigator, Pusen Wang, Principal Investigator, Shenzhen Third People's Hospital
Other Study IDs: SZSPH-LT-mNGS
Record Dates: First submitted 2023-12-26; First posted 2024-01-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid, blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- donor-mNGS-testing group: Organ donors are treated with mNGS testing before organ donation
  Interventions: Diagnostic Test: mNGS
- donor-non-mNGS-testing group: Organ donors are not treated with mNGS testing before organ donation

INTERVENTIONS:
Diagnostic Test: mNGS — metagenomics next generation sequencing
  Groups: donor-mNGS-testing group

SUMMARY:
Liver transplantation is the most efficacious treatment for end-stage liver disease; however, postoperative infection remains a major complication and leading cause of recipient mortality. Specifically, infections originating from donors, particularly those caused by multidrug-resistant bacteria, can significantly impact the prognosis of liver transplant recipients. Theoretically, implementing targeted antimicrobial therapy for donors prior to organ donation could reduce the likelihood of pathogen transmission with the transplanted organ, thereby potentially decreasing the incidence of post-transplant infections from donor sources and improving recipient outcomes. Nevertheless, there is currently a dearth of high-quality prospective studies in this domain. Our previous investigation (Front Microbiol. 2022 Jul 1;13:919363) demonstrated that second-generation metagenomic sequencing (mNGS) technology holds substantial value in expeditious pathogen screening following liver transplantation. Prompt implementation of targeted treatment based on microbiological findings has shown potential to enhance outcomes for select recipients. Therefore, this study aims to provide tailored treatment for donors based on microbiological examination results (including mNGS detection and culture results), analyze corresponding data regarding recipient infection occurrence and prognosis, and explore the impact of mNGS-guided donor antimicrobial therapy on perioperative infection rates among liver transplant recipients.

DETAILED DESCRIPTION:
Liver transplantation has been established as a highly effective treatment for end-stage liver disease, with continuous advancements in surgical techniques and immunosuppressive regimens significantly improving success rates and long-term survival for recipients. Despite these strides, postoperative challenges persist, with infections remaining a major complication and a leading cause of recipient mortality. Pathogens typically arise from the recipient's lungs, intestines, or other sites, yet donor-derived infections (DDIs), particularly those involving multidrug-resistant organisms, pose a substantial threat to transplant recipients' prognosis, prompting increased attention from liver transplant surgeons. Conventional microbial culture, with its lower positivity rate compared to metagenomic next-generation sequencing (mNGS), exhibits a limited ability to guide clinically targeted anti-infective treatment. Hence, the rapid and accurate identification of pathogens, coupled with early targeted anti-infective treatment, is pivotal for effective post-transplant infection management and DDI prevention. Theoretically, preemptive identification of microbiological diagnoses before organ donation, followed by targeted anti-infective treatment for the donor, holds the potential to diminish the risk of pathogens entering the recipient's body with the donated organ. This reduction may subsequently decrease the risk of post-transplant recipient infection originating from the donor, ultimately enhancing the recipient's prognosis. However, as of now, there is a dearth of relevant clinical research on this topic. Notably, our transplantation center employs mNGS to screen both donor and recipient pathogens, a method progressively gaining widespread clinical application. Through a comprehensive analysis of results from both detection methods, we implement targeted anti-infective treatment for both donors and recipients. Consequently, by analyzing cases of liver transplantation and their corresponding donor cases at our center, this study aims to investigate the impact of donor anti-infective treatment guided by mNGS microbiological diagnosis on the incidence of perioperative infections in recipients undergoing liver transplantation. The analysis encompasses the occurrence of infections, results of microbiological examinations, and the formulation of corresponding anti-infective treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Recipient age >18 years;
* Clinical diagnosis of infection in the donor with administered anti-infective treatment;
* Complete clinical data for both the donor and recipient.

Exclusion Criteria:

* Recipient age <18 years;
* Presence of surgery-related factors leading to death or infection, such as intraoperative cardiac arrest resulting in postoperative death, intraoperative bleeding exceeding 2000ml, postoperative complications like intestinal or bile leakage, graft dysfunction, or small liver syndrome;
* Incomplete clinical data for the donor or recipient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Infection | The study focused on the incidence of infection and the postoperative prognosis of transplant recipients within 30 days
  The diagnosis of infection relies on a comprehensive assessment of clinical manifestations, microbiological test results, imaging examinations, and related laboratory tests. In our study, this diagnosis was established by a team of infectious disease specialists and organ transplant physicians. Donor-derived infection occurs when pathogens present in the donor's body post-organ procurement lead to the recipient contracting an infection with the same pathogens during the organ transplantation process.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhao, Dr., Principal Investigator — Shenzhen Third People's Hospital
Locations (1):
- Shenzhen Third People's Hospital, Shenzhen, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No